CLINICAL TRIAL: NCT06031116
Title: Efficacy of Ceramic Soft Tissue Trimming Bur Versus Conventional Scalpel Technique in Ginigival Depigmentation Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sally Nassar, Dentist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ceramic v blade depigmentation
Record Dates: First submitted 2022-12-19; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: split mouth (dental arches)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ceramic soft tissue bur (Experimental): Eight dental arches were treated by ceramic soft tissue bur
  Interventions: Procedure: depigmentation
- scalpel (Active Comparator): Eight dental arches were treated by conventional scalpel technique
  Interventions: Procedure: depigmentation

INTERVENTIONS:
Procedure: depigmentation — gingival depigmentation

SUMMARY:
the investigator compares the clinical outcomes and pain levels after gingival depigmentation by ceramic soft tissue bur vs scalpel surgery

DETAILED DESCRIPTION:
This clinical study will be carried out to compare the efficacy of ceramic soft tissue trimming bur versus the conventional surgical scraping technique in the management of gingival hyperpigmentation.

This study will be conducted to assess:

Primary objectives:

1. Clinical outcome of the gingival depigmentation procedure.
2. Assessment of postoperative pain using the visual analogue scale.
3. Patients' satisfaction will be assessed using the patient satisfaction questionnaire (short-form, PSQ-18) and the global aesthetic improvement scale.

Secondary objectives:

1. Operating time.
2. Wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Males and females within age range of 20-50 years.
* Systemic (medically) free individuals.
* Gingival pigmentation score > 3 on Hedin melanin index15.
* Patients with good oral hygiene.
* Patients with thick gingival phenotype.

Exclusion Criteria:

* Smokers.
* Teeth with compromised periodontium.
* Pregnant and lactating females.
* The vulnerable group: patients with mental or physical disabilities.
* Medications that cause gingival pigmentation.
* Pathologies that cause gingival pigmentation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
clinical outcomes of depigmentation procedure | 3 month postoperative
  dummet oral pigmentation index ( DOPI): 1= pink no pigmentation (better) 4= deep brown (worse) Melanin index (MI):1= isolated pigment (better), 4= long continous ribbon (worse). reported by visual inspection.
patient satisfaction | 3 months postoperative
  global aesthetic improvement scale 5 point likert scale 1= excellent improvement 5= worsened. patient reported outcome.
  a score from 1 to 5, 1 being better
Percieved pain | 7 days
  postoperative pain will be assessed using visual analoque scale (VAS): 1= being the least pain and 10= being the most severe

SECONDARY OUTCOMES:
operating time | during surgery
  time taken from the beginning of the procedure to its end by stopwatch
Wound healing | 7 days postoperative
  1. Complete reepithelialization
  2. Incomplete reepithelialization
  3. ulcer
  4. tissue defect or necrosis Dummet 1966

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine El sayed, Phd, Study Director — Ain Shams University; Hala Abu elela, Phd, Study Chair — Ain Shams University; Sally Nassar, Bds, Principal Investigator — Ain Shams University
Locations (1):
- Ainshams university, Cairo, Cairo Governorate, Egypt